CLINICAL TRIAL: NCT05438771
Title: The Effects of Ankaferd Hemostat on Preventing Oral Mucositis in Colorectal Cancer Patients Receiving Chemotherapy
Brief Title: The Effects of Ankaferd Blood Stopper
Acronym: ABS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Uludag University (Other)
Responsible Party: Principal Investigator, Yasemin Karacan, Principal investigator, Uludag University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Bursa Uludag University
Record Dates: First submitted 2021-08-09; First posted 2022-06-30 (Actual); Last update posted 2023-06-01 (Actual); Status verified 2023-05

CONDITIONS: Colon Cancer; Oral Mucositis; Nurse's Role; Chemotherapy Effect
Keywords: Colorectal cancer,; Oral Mukozit; Ankaferd Blood Stopper
MeSH Terms: conditions — Colonic Neoplasms; Stomatitis; Colorectal Neoplasms | interventions — ankaferd blood stopper; Toothbrushing; Bicarbonates

STUDY DESIGN:
Intervention Model Description: The study was designed as a randomized controlled experimental study on patients newly diagnosed with colorectal cancer who would receive the first course of FOLFOX combination chemotherapy.
Who Masked: Participant, Care Provider
Masking Description: Which patients would be assigned to the study or control group was determined with the support of a person who was independent of the study and had no knowledge of the research. This person, who had no knowledge about the research, was asked to specify a number, and in the next process, patients were assigned to the study or control group depending on whether the random number was even or odd. Study and control group patients were first evaluated in terms of inclusion criteria. The Consolidated Reporting Trials (CONSORT) diagram was used to randomize patients. The use of the consort diagram has been used to greatly improve the conduct and reporting of randomized controlled trials and to allow the study to be included in future meta-analyses.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bicarbonate (Active Comparator): 1.Correct method of brush Platelet value suitable for tooth brushing Feature of toothbrush (soft, nylon bristled, rounded tip, standard size) Fluoride toothpaste, its amount and use in dry brushes In toothbrush 45 degree, the contact of the bristles with the gums, 4 times contact with the inner, outer, chewing surface, tongue cleaning The benefits of correct brushing (preventing dental plaque and gingival recession, etc.) Importance of brushing teeth twice a day (breakfast and after dinner) Preparation of mouth wash Boiled and cooled water at 100°C Putting 5 measures of boiled and cooled water in a teacup with the 20 ml measuring cup provided.
  Adding 1 teaspoon (6 g) of sodium bicarbonate to water Making a mouthwash Teaching how to gargle with 20 ml of bicarbonate 4 times a day at 6-hour intervals and being asked to spit it out without swallowing,
  Interventions: Other: Bicarbonate
- Ankaferd Blood Stopper (Experimental): Correct method of brush Preparation of the mouthwash Boiled and cooled water at 100°C Putting 4 ml of water in the 5 ml measuring cup given to the patient Putting Ankaferd Blood Stopper on the remaining 1 ml portion of the 5 ml beaker Giving information about making and using mouthwash Use on an empty stomach 2 hours before meals in the morning and at least 2 hours after dinner After rinsing your mouth thoroughly with a mouthwash containing 5 ml of Ankaferd Blood Stopper prepared 2 times a day, you can swallow the solution in your mouth.
  It is said that there is a solution-related discoloration in the mouth and teeth, but that it will return to its original state after tooth brushing.
  Interventions: Combination Product: Ankaferd Blood Stopper

INTERVENTIONS:
Combination Product: Ankaferd Blood Stopper — mouth wash
  Other Names: brushing teeth
  Arms: Ankaferd Blood Stopper
Other: Bicarbonate — mouth wash
  Other Names: brushing teeth
  Arms: Bicarbonate

SUMMARY:
The purpose of oral care is to reduce the effect of oral pathological microbial flora and to prevent infection, pain, and bleeding associated with cancer treatment. New agents are introduced each day to be used in the prevention and treatment of mucositis in cancer treatment. One of those agents is the Ankaferd Hemostat. Ankaferd Hemostat has pleiotropic effects and anti-infective characteristics in tissue healing. The aim of this study is to evaluate the effectiveness of the Ankaferd Hemostat in the prevention of oral mucositis due to chemotherapy in adult patients diagnosed with colorectal cancer.

The study was designed as a randomized controlled experimental study to be conducted with patients who are recently diagnosed with colorectal cancer and will receive the first course of chemotherapyd. The data were collected using the Performance Score and the Oral Mucositis Evaluation Scale.

DETAILED DESCRIPTION:
In patients with colorectal cancer, it is important to perform symptom management dynamically as well as specific treatments for cancer. It is extremely important for healthcare professionals to know the approaches that can be recommended to patients in the management of treatment and disease-related symptoms, in order to prevent problems that may develop in patients due to the severity of symptoms. Controlling the symptoms will increase the patient's functional capacity and quality of life.

Oral mucositis is one of the common toxic effects of chemotherapy. Pain due to mucositis causes anorexia-dysphagia development and malnutrition. As a result, systemic infections can develop, dose reduction in chemotherapy courses, increase in cost and prolongation of hospital stay. Looking at the literature, chloroxidine, glutamine, palifermin was used to prevent the development of mucositis during 5-Fu-based therapy for colon cancer. Solutions such as bicarbonate were used. Although it was determined in these studies to prevent the development of oral mucositis, the incidence of mucositis is still high. Therefore, the search for new treatments and applications to prevent mucositis continues. Ankaferd Hemostat is a herbal product used as a hemostatic agent in traditional Turkish medicine. Ankaferd Hemostat affects endothelium, blood cells, angiogenesis, cellular reproduction and vascular dynamics and stimulates mediators that lead to rapidly progressive wound healing. In addition to these, the anti-inflammatory, antimicrobial, antifungal and antioxidative effects of Ankaferd Hemostat are mentioned in the literature. In order to determine the effectiveness of Ankaferd Hemostat application in chemotherapy-induced oral mucositis in adult patients, there is a single study conducted on 20 patients with mucositis grade 2-3 with hematological malignancy. While it is stated in the literature that the healing time of mucositis is the week after 7-14 days, it was seen that this decreased to 6.6 (3-10) days in the study conducted by Atay.

In another study conducted in the field of dentistry, the effectiveness of Ankaferd Hemostat in preventing the development of oroantral fistula was evaluated. In a study comparing the use of Platelet Rich Plasma (PRP) in one arm and Ankaferd Hemostat in the other arm, it was found that the antibacterial effect was more prominent in the Ankaferd Hemostat arm and the results of edema, bleeding and infection were similar in both arms .

ELIGIBILITY:
Inclusion Criteria:

* between the ages of 18-75
* At least primary school graduate
* No communication problems
* No mouth sores/mucositis (Mucositis stage=0)
* Having been diagnosed with colorectal cancer
* To receive Folfox (5-Fluorouracil, oxalplatin, folinic acid) combination therapy as first-line therapy Not having received chemotherapy or radiotherapy with any other diagnosis before
* Agreeing to participate in the study
* ECOG performance status 0-2

Exclusion Criteria:

Don't be a denture

* Having an oral herpes simplex lesion
* Smoking
* Using Glutemine Research
* Receiving G-CSF support
* Having a physical disability that prevents them from using the right brushing technique

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2023-06-02 (Estimated); Study Completion 2023-06-02 (Estimated)

PRIMARY OUTCOMES:
Personal Information Form | day 1
  This form, which was created as a result of literature review by the researchers at the beginning of the study, was prepared for both the study and control group patients included in the sample. It consists of 12 questions including brushing habits and the person responsible for its care) and health status and habits (having another chronic disease, smoking and alcohol use).
ECOG Performance Score (Eastern Cooperative Oncology Group) | Up to Day 15
  The Eastern Cooperative Oncology Group (ECOG) performance scale, also known as the WHO or Zubrod performance score, was developed in 1960. On the ECOG Performance scale, 0 means normal health and 5 means death. Low scores indicate good general condition, while high scores indicate poor prognosis. '0' Normal. Can maintain normal activity before the disease, '1' Can continue his daily life with bearable tumor findings, '2', Has disturbing tumor findings but spends more than 50% of his time out of bed, '3' Is severely disturbed and spends % of his time It is evaluated as '4' Being in a very uncomfortable condition and spending all his time tied to the bed, '5' Dead, who had to stay more than 50 of them tied to the bed.
Oral Care Control Chart | Up to Day 15
  This form was developed by the researchers in order to ensure that patients' oral care intervals, tooth brushing and mouthwash are made and to prevent them from being forgotten. It was used to record the oral care performed by the patients in the intervention and control groups during the follow-up period. The form is a checklist to be filled by clicking after oral care.

SECONDARY OUTCOMES:
Number of participants with abnormal laboratory test results | Up to Day 15
  hemoglobin, hematocrit, neutrofil, body mass index

OTHER OUTCOMES:
World Health Organization (WHO) Oral Mucositis Evaluation | Up to Day 15
  It is a grading system developed by WHO according to the clinical appearance and functional status of mucositis. WHO evaluates oral mucositis (OM) as subjective (patient-described pain), objective (presence of erythema and ulcerations) and functional (ability to consume liquid/solid foods by mouth or inability to eat anything). OM grade 0 (normal), grade 1 [mild focal changes (erythematous areas) no pain and tenderness yet, can be fed orally], grade 2 (painless ulcers, erythema, mild pain sensation), grade 3 (painful erythema, edema or ulcers) (depth >2 mm and less than half of the mucosa) no bleeding, can only be fed orally with liquid diet) and grade 4 (erythema, edema or ulcers (more than half the mucosa), severe pain, bleeding, no nutrition, parenteral and enteral nutrition support may be required)
patient education | Up to Day 15
  Patients were informed about the precaution of oral hygiene. The patients were instructed to brush their teeth at least twice a day, morning and evening. Toothbrushes with soft nylon bristles with rounded ends were given to the patients. Modified Stillman method for tooth brushing was taught. The bristle ends of the brush should be placed in the apical direction, against the cervical part of the teeth and partially against the adjacent gingiva (it should be activated with a back-and-forth motion at least 4 times on each tooth at an angle of 450 and simultaneously move it in the coronal direction (from bottom to top, from right to left). announced.

CONTACTS AND LOCATIONS:
Overall Officials: Hicran Yıldız, Study Director — Hicran Yıldız
Locations (1):
- Bursa Uludag University, Bursa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
I can share after the work is done

REFERENCES:
- [Result] Elad S. The MASCC/ISOO Mucositis Guidelines 2019 Update: introduction to the first set of articles. Support Care Cancer. 2019 Oct;27(10):3929-3931. doi: 10.1007/s00520-019-04895-x. Epub 2019 Jul 8. No abstract available. PMID 31286226
- [Result] Djuric M, Hillier-Kolarov V, Belic A, Jankovic L. Mucositis prevention by improved dental care in acute leukemia patients. Support Care Cancer. 2006 Feb;14(2):137-46. doi: 10.1007/s00520-005-0867-7. Epub 2005 Jul 22. PMID 16041502
- [Result] Dekker E, Tanis PJ, Vleugels JLA, Kasi PM, Wallace MB. Colorectal cancer. Lancet. 2019 Oct 19;394(10207):1467-1480. doi: 10.1016/S0140-6736(19)32319-0. PMID 31631858
- [Result] Goker H, Haznedaroglu IC, Ercetin S, Kirazli S, Akman U, Ozturk Y, Firat HC. Haemostatic actions of the folkloric medicinal plant extract Ankaferd Blood Stopper. J Int Med Res. 2008 Jan-Feb;36(1):163-70. doi: 10.1177/147323000803600121. PMID 18304416
- [Result] Orhan I, Dogan R, Soylu E, Aksoy F, Veyseller B, Ozturan O, Esrefoglu M, Aydin MS. Histopathological evaluation of Ankaferd blood stopper use in the rabbit septoplasty model. Int J Pediatr Otorhinolaryngol. 2015 Mar;79(3):305-9. doi: 10.1016/j.ijporl.2014.11.015. Epub 2014 Dec 15. PMID 25596649
- [Result] Saito H, Watanabe Y, Sato K, Ikawa H, Yoshida Y, Katakura A, Takayama S, Sato M. Effects of professional oral health care on reducing the risk of chemotherapy-induced oral mucositis. Support Care Cancer. 2014 Nov;22(11):2935-40. doi: 10.1007/s00520-014-2282-4. Epub 2014 May 23. PMID 24854326
- [Result] Sonis ST. Mucositis as a biological process: a new hypothesis for the development of chemotherapy-induced stomatotoxicity. Oral Oncol. 1998 Jan;34(1):39-43. doi: 10.1016/s1368-8375(97)00053-5. PMID 9659518
- [Derived] Karacan Y, Yildiz H, Evrensel T, Haznedaroglu IC. The effects of Ankaferd hemostat on preventing oral mucositis in colorectal cancer patients receiving chemotherapy. Support Care Cancer. 2023 Jun 8;31(7):385. doi: 10.1007/s00520-023-07856-7. PMID 37289263

DOCUMENTS (1):
  • Study Protocol (2022-06-06): https://cdn.clinicaltrials.gov/large-docs/71/NCT05438771/Prot_000.pdf